CLINICAL TRIAL: NCT06061250
Title: Effects of Preoperative Gum Chewing on Postoperative Sore Throat After Double-lumen Endobronchial Tube Intubation: A Randomized Controlled Trial
Brief Title: Effect of Gum Chewing on Sore Throat After Double-lumen Tube Intubation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has not commenced due to medical staff strikes and staffing shortages.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, PhD, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2308-119-1459
Record Dates: First submitted 2023-09-21; First posted 2023-09-29 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Thoracic Surgery, Video-Assisted; Chewing Gum; Pharyngeal Diseases
MeSH Terms: conditions — Pharyngeal Diseases

STUDY DESIGN:
Intervention Model Description: Two separate groups of patients will undergo same anesthetic procedure, except for chewing a gum for 2 minutes or swallowing saliva twice 10 minutes before the induction of anesthesia.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gum group (Experimental): This group of patients will receive a piece of Xylitol gum (LOTTE WELLFOOD, Korea) 10 minutes before induction of anesthesia. Patients will chew it for 2 minutes and spit out. Other anesthetic care will follow routine protocol of the hospital.
  Interventions: Dietary Supplement: Chewing a piece of gum (Xylitol gum, LOTTE WELLFOOD, Korea) before induction of anesthesia
- Control group (No Intervention): This group of patients will instructed to swallow their saliva twice 10 minutes before induction of anesthesia. Other anesthetic care will follow routine protocol of the hospital.

INTERVENTIONS:
Dietary Supplement: Chewing a piece of gum (Xylitol gum, LOTTE WELLFOOD, Korea) before induction of anesthesia — To replicate Xylitol chewing gum, which has been shown to reduce postoperative sore throat in previous studies of single-lumen endotracheal tubes and supraglottic airways, the investigators will use a commercially available gum from South Korea.
  Arms: Gum group

SUMMARY:
Patients undergoing video-assisted thoracoscopic surgery requiring double-lumen tube intubation are randomized into two groups; gum group and control group. In the gum group, patients are instructed to chew gum for 2 minutes, approximately 10 minutes before induction of anesthesia. Patients in the control group are instructed to swallow saliva twice. Postoperative sore throat and hoarseness are assessed 30 minutes after recovery room admission, and at 2 and 24 hours after extubation.

DETAILED DESCRIPTION:
Patients scheduled for video-assisted thoracoscopic surgery requiring double-lumen tube intubation and who agree to participate in the study are randomized to the gum chewing group and the control group. All clinical procedures are identical in both groups except for preoperative gum chewing. The gum chewing group chew gum for approximately 2 minutes, 10 minutes before induction of anesthesia. The control group do not chew gum and be induced to swallow saliva twice at the same time point. All patients are endotracheally intubated with a double-lumen tube using video laryngoscopy to provide unilateral pulmonary ventilation. Extubation is performed according to routine procedures, and the tube is assessed with whether there are blood stains at extubation. At 30 minutes in the recovery room and at 2 hours and 24 hours after extubation, the patient's sore throat is assessed for presence and intensity assessed by a 11-point numerical pain scale (minimal value 0 representing absence of pain, maximal value 10 representing the worst possible pain). Hoarseness at the same time points is also assessed for presence and severity. The presence of intubation-related complications (aspiration pneumonia) is assessed as a safety measure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-75 years undergoing routine video-assisted thoracoscopic surgery scheduled for double-lumen tube intubation
* Patients who are able to provide written informed consent to participate in the study and understand the procedures of this study
* American Society of Anesthesiologists physical status classification (ASA physical status classification) grade 1-2

Exclusion Criteria:

* Patients who have not consented to the study
* American Society of Anesthesiologists physical status classification (ASA physical status classification) grade 3-4
* Patients with poor dental health that limits chewing gum or tracheal intubation
* Patients who are expected to be difficult to intubate
* Patients with a history of aspiration pneumonia
* Patients being treated for chronic laryngitis, chronic bronchitis, asthma, reflux esophagitis
* Patients with a history of smoking within the past week
* Patients who have difficulty communicating or carrying out gum chewing and spitting instructions
* Patients with hypersensitivity to Xylitol gum ingredients
* Patients taking narcotic analgesics, antidepressants, and anticonvulsants for chronic pain
* Patients requiring endotracheal intubation or intensive care unit treatment after surgery
* Patients who, in the opinion of the investigator or study staff, are not appropriate candidates for this study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-24 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative sore throat at 24 hours after extubation | 24 hours after extubation
  Incidence of postoperative sore throat at 24 hours after extubation, described as percentage of patients with sore throat out of all patients in the same group.

SECONDARY OUTCOMES:
Intensity of postoperative sore throat at 24 hours after extubation | 24 hours after extubation
  Intensity of postoperative sore throat at 24 hours after extubation, assessed with 11-point numeric rating scale (minimal value 0 representing absence of pain, maximal value 10 representing the worst possible pain).
Incidence of postoperative sore throat at 30 minutes in recovery room and 2 hours after extubation | 30 minutes in recovery room and 2 hours after extubation
  Incidence of postoperative sore throat at 30 minutes in recovery room and 2 hours after extubation, described as percentage of patients with sore throat out of all patients in the same group.
Intensity of postoperative sore throat at 30 minutes in recovery room and 2 hours after extubation | 30 minutes in recovery room and 2 hours after extubation
  Intensity of postoperative sore throat at 30 minutes in recovery room and 2 hours after extubation, assessed with 11-point numeric rating scale (minimal value 0 representing absence of pain, maximal value 10 representing the worst possible pain).
Incidence of hoarseness at 30 minutes in recovery room, and at 2 and 24 hours after extubation | At 30 minutes in recovery room, and at 2 and 24 hours after extubation
  Incidence of hoarseness at 30 minutes in recovery room, and at 2 and 24 hours after extubation, described as percentage of patients with hoarseness out of all patients in the same group.
Intensity of hoarseness at 30 minutes in recovery room, and at 2 and 24 hours after extubation | At 30 minutes in recovery room, and at 2 and 24 hours after extubation
  Intensity of hoarseness at 30 minutes in recovery room, and at 2 and 24 hours after extubation, assessed with 4-step scale (none, mild, moderate, and severe).